CLINICAL TRIAL: NCT00790439
Title: Open Randomized Multi-Center Study to Evaluate Safety and Efficacy of Low Molecular Weight Sulfated Dextran (LMW-SD) in Islet Transplantation After Kidney Transplantation (CIT-01B)
Brief Title: Safety and Effectiveness of Low Molecular Weight Sulfated Dextran in Islet Transplantation After Kidney Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to funding limitations
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-01B; CIT-01B
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Insulin dependence
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Heparin; Mycophenolic Acid; Sirolimus; Tacrolimus; Cyclosporine; Cyclosporins; Daclizumab; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMW-SD (Experimental): 18 participants randomized to immunosuppression with Low Molecular Weight Sulfated Dextran (LMW-SD)
  Interventions: Drug: Low Molecular Weight Sulfated Dextran; Drug: Mycophenolate Mofetil; Drug: Sirolimus; Drug: Tacrolimus; Drug: Cyclosporine; Drug: Daclizumab; Drug: Basiliximab; Biological: Allogeneic Pancreatic Islet Cells
- Control Group, Standard of Care (Active Comparator): 18 participants randomized to immunosuppression without Low Molecular Weight Sulfated Dextran (LMW-SD)
  Interventions: Drug: Heparin; Drug: Mycophenolate Mofetil; Drug: Sirolimus; Drug: Tacrolimus; Drug: Cyclosporine; Drug: Daclizumab; Drug: Basiliximab; Biological: Allogeneic Pancreatic Islet Cells

INTERVENTIONS:
Drug: Low Molecular Weight Sulfated Dextran — Inhibitor of instant blood-mediated inflammatory reaction
  Other Names: LMW-SD
  Arms: LMW-SD
Drug: Heparin — Anticoagulant
  Other Names: Heparin Sodium
  Arms: Control Group, Standard of Care
Drug: Mycophenolate Mofetil — Cell proliferation inhibitor, Transplantation (immunosuppressive)
  Other Names: MMF; Mycophenolate; Mycophenolic Acid; CellCept
Drug: Sirolimus — Cell proliferation inhibitor, immunologic (immunosuppressive)
  Other Names: Rapamune
Drug: Tacrolimus — Calcineurin inhibitor
  Other Names: Hecoria
Drug: Cyclosporine — Calcineurin inhibitor, immunosuppressant
  Other Names: Ciclosporin; GENGRAF® Capsules
Drug: Daclizumab — Monoclonal IL-2 receptor blocker
Drug: Basiliximab — Monoclonal IL-2 receptor blocker
  Other Names: Simulect ®
Biological: Allogeneic Pancreatic Islet Cells

SUMMARY:
Type 1 diabetes mellitus (T1D) is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to assess the safety and effectiveness of low molecular weight sulfated dextran (LMW-SD) on post-transplant islet function in people with T1D who have responded to intensive insulin therapy and have received kidney transplants. This study is taking place in Uppsala and Stockholm, Sweden, and Oslo, Norway.

DETAILED DESCRIPTION:
T1D is commonly treated with the administration of insulin, either by multiple insulin injections or by a continuous supply of insulin through a wearable pump. Insulin therapy allows long-term survival in individuals with T1D; however, it does not guarantee constant normal blood sugar control. Because of this, long-term type 1 diabetic survivors often develop vascular complications, such as diabetic retinopathy, an eye disease that can cause poor vision and blindness, and diabetic nephropathy, a kidney disease that can lead to kidney failure and thus kidney transplant. Some individuals with T1D develop hypoglycemia unawareness, a life-threatening condition that is not easily treatable with medication and is characterized by reduced or absent warning signals for hypoglycemia. For such individuals, pancreas or pancreatic islet transplantation are possible treatment options. Rejection of these islets by the recipient's immune system, however, can make the treatment ineffective. An immune response known as instant blood-mediated inflammatory reaction (IBMIR) results in the disruption of islet integrity and islet loss within an hour of transplantation. LMW-SD inhibits IBMIR by preventing the cascade that triggers it, when combined with pancreatic islets. The purpose of this study is to determine the safety and efficacy of LMW-SD improving the outcome of islet transplantation by preventing IBMIR.

Once a preparation of islets becomes available, participants will be randomly assigned to either the low molecular weight sulfated dextran (LMW-SD) Arm or to the Control Group/Standard of Care Arm. Participants in the LMW-SD Arm will receive LMW-SD before, with and for 5 hours after islet transplantation. Participants in the Control Group will receive heparin with the islet transplantation. All participants will also receive the oral medications, mycophenolate mofetil or sirolimus and tacrolimus or cyclosporine throughout the study. In addition, they will receive either intravenous daclizumab on the day of islet transplantation and at Week 2, 4, 6, and 8 or intravenous basiliximab on the day of islet transplantation and on Day 4. The islet transplantation will occur at the hospital and will be given via the portal vein. All participants will be eligible to receive second and third islet transplantation(s) if previous transplants fail. After each islet transplantation, study visits will occur on Days 1, 3, 7, 14, 21, 28, 75, and Months 6 and 12. At these visits, physical exams and blood collection will occur. At some visits urine collection will also occur.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to provide written informed consent and comply with study procedures
* Clinical history compatible with T1D and onset of disease at less than 40 years of age and insulin dependence for more than (>) 5 years at the time of enrollment; AND the sum of subject age and insulin-dependent diabetes duration is >=28
* Absent stimulated C-peptide (less than 0.3 ng/mL) 60 and 90 minutes post-mixed-meal tolerance test (MMTT)
* Subjects >6 months post renal (kidney) transplant, currently taking or willing to switch to appropriate maintenance immunosuppression
* Stable renal function and free of rejection for >=3 months prior to islet transplantation
* Standard medical treatment for >=3 months under the care of an experienced diabetologist and at the end of this period has had at least 1 severe hypoglycemic event OR a hemoglobin A1C (HbA1c) >7.2% OR reduced awareness of hypoglycemia manifest by a Clark score of >=4 in the last year prior to study entry

Exclusion Criteria:

* Known immunoglobulin E (IgE) mediated allergy to antibiotics used in islet culture medium
* Known hypersensitivity to dextran
* Measured glomerular filtration rate (GFR) using Iothalmate, 51Cr-EDTA, 99-technetium-DPTA, or iohexol of less than 40ml/min/1.73 m^2
* Proteinuria (albuminuria greater than 500 mg in 24 hours) of new onset since kidney transplantation
* Other (non-kidney) organ transplants except prior failed pancreatic graft
* Body mass index (BMI) >30 kg/m^2
* Insulin requirement of >1.0 IU/kg/day
* Consistently abnormal liver function tests (aspartate aminotransferase(AST), alanine aminotransferase (ALT),alkaline phosphatase, or total bilirubin) of greater than 1.5 times the upper limit of normal for two consecutive measurements that are >2 weeks apart
* Untreated proliferative diabetic retinopathy
* History of hypercoagulability disorder or coagulopathy or International Normalized Ratio(INR) that is >1.5
* Activated Protein C Resistance (APC-R)
* Evidence by serologies and PCR of acute or chronic active Epstein-Barr Virus (EBV) infection OR no evidence by EBV serologies of prior EBV exposure
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known history of severe co-existing cardiac disease, characterized by any one of the following conditions:

  1. Recent myocardial infarction (<=6 months)
  2. Evidence of ischemia on functional cardiac exam <=last year
  3. Left ventricular ejection fraction <30%
* Active infections, unless treatment is not judged necessary by the investigators(including but not limited to mild skin and nail fungal infections)
* Active infection including hepatitis B, hepatitis C,human immunodeficiency virus (HIV), or pulmonary tuberculosis
* Subjects with active peptic ulcer disease, symptomatic gallstones or portal hypertension
* Acute or chronic pancreatitis
* Subjects who are pregnant or breastfeeding, or who intend to become pregnant
* Sexually-active females who are not: a) post-menopausal, b) surgically sterile, or c) using an acceptable method of contraception: oral contraceptives, Norplant, Depo-Provera, and barrier devices combined with spermicidal gel are acceptable; condoms used alone are not acceptable.
* Active alcohol or substance abuse
* Evidence of high-level sensitization (Panel Reactive Antibodies (PRA) >50%) or positive cross match or the known presence of anti-donor HLA class I antibodies
* Treatment with any anti-diabetic medication, other than insulin, <=4 weeks of enrollment
* Use of any investigational agents <=4 weeks of enrollment
* Receipt of live attenuated vaccine(s) <=2 months of enrollment
* Subjects with any condition or circumstance that in the opinion of the investigator would make it unsafe to undergo an islet transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Level of Stimulated C-peptide at 90-minutes in Response to a Mixed-Meal Tolerance Test (MMTT) | 75 days following the first islet transplantation

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events Related to the Islet Transplantation Procedure | 75 days and 365 days following the first islet transplantation
Incidence and Severity of Adverse Events Related to the Immunosuppression | 75 days and 365 days following the first islet transplantation
Incidence of Immune Sensitization Defined by Detecting Anti-HLA (Human Leukocyte Antigen) Antibodies not present prior to transplantation | 75 days and 365 days following the first islet transplantation
  Defined by detecting anti-HLA (Human Leukocyte Antigen) antibodies not present prior to transplantation
Incidence of a Change in the Immunosuppression Drug Regimen | 75 days and 365 days following the first islet transplantation
Incidence of Worsening Retinopathy | 365 days following the first islet transplantation
  As assessed by change in retinal photography from pre-transplant to 365 days following the first islet transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Olle Korsgren, MD, Principal Investigator — Department of Oncology, Radiology, and Clinical Immunology, Rudbeck Laboratory, Uppsala University Hospital

REFERENCES:
- See also: Click here for the Clinical Islet Transplantation Consortium Web site — http://www.CITISletstudy.org
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/Pages/default.aspx